CLINICAL TRIAL: NCT04785859
Title: Multiparametric Prediction of the Risk of Moderate-severe Bronchopulmonary Dysplasia in Neonates Born Before 30 Weeks of Gestation
Brief Title: Multiparametric Bronchopulmonary Prediction
Acronym: PARADYS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andaluz Health Service (Other Government)
Collaborators: University of Cadiz (Other); European Society of Pediatric and Neonatal Intensive Care (Unknown)
Responsible Party: Principal Investigator, Almudena Alonso Ojembarrena, Dr., Andaluz Health Service
Other Study IDs: NEO-LUS-20-01
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Lung ultrasound, NICU, Premature, Proteomics
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal aspirates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate-severe bronchopulmonary dysplasia: Neonates of less than 30 weeks´ gestation, born at any of the study centers, or transferred from other centers in the first 24 hours of life, with the diagnosis of moderate-severe bronchopulmonary dysplasia at 36 weeks' postmenstrual age.
  Interventions: Diagnostic Test: BPD prediction
- no moderate-severe bronchopulmonary dysplasia: Neonates of less than 30 weeks´ gestation, born at any of the study centers, or transferred from other centers in the first 24 hours of life, without the diagnosis of moderate-severe bronchopulmonary dysplasia at 36 weeks' postmenstrual age.
  Interventions: Diagnostic Test: BPD prediction

INTERVENTIONS:
Diagnostic Test: BPD prediction — The following lung ultrasounds will be performed on the patients included in the study: first 24 hours of life, 3rd day of life (DOL) and 7th DOL. At one week of life detection of proteins in nasopharyngeal aspirates will be performed. During the first week of life, an echocardiography will be performed in all patients to evaluate the possibility of a patent ductus arteriosus and its hemodynamic significance.
  In the first 20 patients who remain intubated at one week of life, tracheal aspirates will be obtained too, to compare protein determination in both aspirates at the same time.

SUMMARY:
INTRODUCTION: Current Neonatology has failed to reduce the incidence of moderate-severe bronchopulmonary dysplasia (BPD). Although multiple models for predicting the risk of dysplasia in preterm infants have been studied, none have been implemented in clinical practice.

OBJECTIVE: To calculate a mathematical model to predict moderate-severe bronchopulmonary dysplasia in newborns before 30 weeks of gestation based on pre and postnatal clinical variables, lung ultrasound images and detection of biomarkers in nasopharyngeal aspirate.

METHODOLOGY: Multicenter case-control study, in which 10 Spanish neonatal intensive care units (NICU) will participate. All participants will undergo a lung ultrasound in the first 24 hours, on the third day of life, at one week and two weeks of life, a nasopharyngeal aspirate at one week of life, and cardiac ultrasound at one week and two weeks of life. It is expected to include 240 patients in 29 months of study among all participating units: 200 for the calculation of the model, and 40 more for its subsequent validation. These will be divided between those with a diagnosis of moderate-severe BPD and those without, and the values of each of the variables described in the methodology section will be compared between the two groups. Those with a significant difference will be entered into a logistic regression model to calculate those that best predict the final diagnosis. With the results of the calculated model, a mobile application will be created with a risk of moderate-severe BPD calculator in this population, for its worldwide distribution.

DETAILED DESCRIPTION:
Type of study: case-control study. Study population: Neonates of less than 30 weeks´ gestation, born at any of the study centers, or transferred from other centers in the first 24 hours of life, during the study period. The participating hospitals will be: Puerta del Mar University Hospital in Cádiz, Basurto University Hospital in Bilbao, Álvaro Cunqueiro University Hospital in Vigo, Doctor Josep Trueta University Hospital in Girona, Clínic University Hospital in Barcelona, León University Hospital, Gregorio Marañón University Hospital in Madrid, German Trias i Pujol Hospital in Barcelona, Miguel Servet Hospital in Zaragoza and Val d'Hebron Hospital in Barcelona.

Study protocol: The following lung ultrasounds will be performed on the patients included in the study: first 24 hours of life, 3rd day of life (DOL) and 7th DOL. At one week of life detection of proteins in nasopharyngeal aspirates will be performed. During the first week of life, an echocardiography will be performed in all patients to evaluate the possibility of a patent ductus arteriosus and its hemodynamic significance.

In the first 20 patients who remain intubated at one week of life, tracheal aspirates will be obtained too, to compare protein determination

ELIGIBILITY:
Inclusion Criteria:

* Neonates of less than 30 weeks´ gestation, born at any of the study centers, or transferred from other centers in the first 24 hours of life, during the study period

Exclusion Criteria:

* Neonates with severe chromosomal abnormalities, or severe congenital anomalies, infants who died prior to 36 weeks´ corrected age, as well as patients whose clinical condition prevents the performance of the study protocol ultrasounds.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates born before 30 weeks' gestation.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
multiparametric moderate-severe BPD prediction | 7 days
  • To assess if LUS and respiratory tract inflammatory parameters in the first week of life of preterm babies born before 30 weeks´ gestation, improves the predictive power of epidemiological and clinical variables for moderate-severe BPD.

SECONDARY OUTCOMES:
respiratory variables prediction by LUS | 7 days
  • To assess the predictive value of LUS in the first week of life in the diagnosis of moderate-severe BPD, the total duration of respiratory support, oxygen therapy and the need for home oxygen therapy.
Diffusion of the models obtained | After 36 weeks' postmenstrual age
  • To create a website with a risk calculator for moderate-severe BPD in preterm infants of less than 30 weeks´ gestation, depending on the data obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta del Mar, Cadiz, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrido-Munoz F, Fernandez-Vega A, Gregorio-Hernandez R, Padin-Fontan M, Heras-Martin ML, Teresa-Palacio M, Alonso-Quintela P, Trujillo-Fagundo A, Perez-Perez A, Pumarada-Prieto M, Montero-Gato J, Aldecoa-Bilbao V, Oulego-Erroz I, Sanchez-Fernandez M, Alonso-Ojembarrena A. Proteomic Analysis of Nasopharyngeal Aspirate Biomarkers for Prematurity-Related Bronchopulmonary Dysplasia. Chest. 2025 Oct;168(4):980-993. doi: 10.1016/j.chest.2025.04.036. Epub 2025 May 12. PMID 40368027